CLINICAL TRIAL: NCT04059237
Title: Pilot Study of a Decision Aid Intervention for Family-building After Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Catherine Benedict, Clinical Associate Professor, Psychiatry and Behavioral Sciences- Medical Psychiatry, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB-52143; VAR0190 (Other: OnCore); IRB-52143 (Other: Stanford IRB); K07CA229186 (NIH)
Record Dates: First submitted 2019-08-14; First posted 2019-08-16 (Actual); Results first posted 2024-04-09 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-03

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Online Decision Aid (Experimental): web-based psychosocial assessment questionnaires will be administered at baseline (T1; pre-intervention) and at one-month (T2) and three-month (T3) follow-up time points.
  Interventions: Behavioral: Web based decision aid intervention

INTERVENTIONS:
Behavioral: Web based decision aid intervention — Decision aid tool (website) to assist young adult female cancer survivors in making decisions and preparing for family-building after cancer.

SUMMARY:
This study tests a web-based decision aid and planning too to help young female cancer survivors manage fertility and family-building issues in post treatment survivorship.

DETAILED DESCRIPTION:
The overall goal of this work is to pilot test a single-arm intervention of a decision aid and planning tool (website) to assist young adult female cancer survivors in making decisions and preparing for family-building after cancer.

Primary Objective: Examine feasibility and acceptability of a decision aid intervention in a single-arm pilot trial.

Secondary Objective: Obtain preliminary effect sizes of the decision aid intervention using a pre-post study design.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Completed cancer treatment known to have gonadotoxic effects (e.g., systemic chemotherapy, surgery affecting reproductive organs or hormone regulation, and/or pelvic radiation)
* Understands verbal and written English
* Desires future children or uncertainty regarding family-building plans
* Access to the Internet and use of a computer, tablet, or smartphone

Exclusion Criteria:

* Currently undergoing cancer treatment excluding long-term adjuvant or maintenance therapies, such as tamoxifen
* Significant physical or mental disability that prevents completion of study activities

Note: Survivors on adjuvant maintenance or endocrine treatment, such as tamoxifen, will not be excluded because clinical guidelines allow treatment delay or hiatus to accommodate fertility preservation, egg extraction for surrogacy, or pregnancy for some patients, and because patients may be interested in alternative family-building options such as surrogacy or adopting.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 102 (Actual)
Dates: Start 2020-01-06 (Actual); Primary Completion 2022-12-11 (Actual); Study Completion 2022-12-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Benedict, Principal Investigator — Stanford University
Locations (1):
- Stanford Cancer Center, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Benedict C, Ford JS, Schapira L, Simon P, Spiegel D, Diefenbach M. Family-building decision aid and planning tool for young adult women after cancer treatment: protocol for preliminary testing of a web-based decision support intervention in a single-arm pilot study. BMJ Open. 2019 Dec 29;9(12):e033630. doi: 10.1136/bmjopen-2019-033630. PMID 31888941

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 102 participants signed informed consent; 98 participants started the study.
Period: Overall Study
Arm/Group | Online Decision Aid
Started | 98
Completed Baseline Assessment | 98
Completed 1-month Assessment | 78
Completed 3-month Assessment | 55
Completed | 55
Not Completed | 43

BASELINE CHARACTERISTICS:
Arm/Group | Online Decision Aid
Number analyzed (Participants) | 98
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.98 (5.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 98
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14
  Not Hispanic or Latino | 84
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 84
  Black | 4
  Asian or Pacific Islander | 6
  Other | 3
  Prefer not to answer | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 98

OUTCOME MEASURES:

1. Primary Outcome: Measure Decision Conflict Scale
Description: The Decisional Conflict Scale (DCS) is a validated survey that assesses personal uncertainty in making healthcare decisions; modifiable factors contributing to uncertainty; and the quality of the decision made. It is reliable and responsive to change, and the most widely used measure of decision-making quality. The survey has 16 questions, with responses on a 5-point scale ranging from "strongly agree" (1) to "strongly disagree" (5). Total scores range from 16 to 80, with higher scores indicating greater uncertainty (worse outcome).
Time Frame: Baseline, 1 month, 3 months
Population: Participants with available data at each respective timepoint
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Online Decision Aid
Number analyzed (Participants) | 98
score on a scale
  Baseline | 52.25 (24.26)
  1 month: number analyzed (Participants) | 78
  1 month | 36.86 (26.03)
  3 months: number analyzed (Participants) | 55
  3 months | 34.55 (16.96)
Statistical Analysis 1: Comparison: Online Decision Aid; Test type: Other; p < 0.001, ANOVA — Repeated measures ANOVA evaluated change in outcome variables across the study time points

2. Secondary Outcome: Fertility Information Needs
Description: This investigator-designed survey assesses perceived information needs about fertility topics such as the risk of infertility; risk of early menopause; options to assess fertility status; options to preserve fertility; and options for alternative family-building. The survey has 5 questions, each answered by a Yes / No response. Yes is scored as 1, and no is scored as 0. Total scores range from 0 to 5, with higher scores indicating greater perceived knowledge.
Time Frame: Baseline, 1 month, 3 months
Population: Participants with available data at each respective timepoint
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Online Decision Aid
Number analyzed (Participants) | 98
score on a scale
  Baseline | 3.39 (1.81)
  1 month: number analyzed (Participants) | 78
  1 month | 2.02 (1.56)
  3 months: number analyzed (Participants) | 55
  3 months | 2.09 (1.67)
Statistical Analysis 1: Comparison: Online Decision Aid; Test type: Other; p < .001, ANOVA — Repeated measures ANOVA evaluated change in outcome variables across the study time points

3. Secondary Outcome: Measure Illness Perceptions Questionnaire-Revised (IPQ-R)
Description: The Illness Perceptions Questionnaire-Revised (IPQ-R) is a survey that assesses cognitive and emotional representations of illness, and is validated in cancer populations. The survey has 28 questions, answered on a 5-point scale ranging from "strongly disagree" (1) to "strongly agree" (5). Mean scores range from 28 to 140, with higher scores indicating worse outcomes. The outcome will be reported as the mean difference from baseline to 1 and 3 months, with standard deviation.
Time Frame: Baseline, 1 month, 3 month
Population: Participants with available data at each respective timepoint
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Online Decision Aid
Number analyzed (Participants) | 98
score on a scale
  Baseline | 85.66 (10.62)
  1 month: number analyzed (Participants) | 78
  1 month | 81.48 (9.94)
  3 months: number analyzed (Participants) | 55
  3 months | 81.64 (10.64)
Statistical Analysis 1: Comparison: Online Decision Aid; Test type: Other; p < 0.001, ANOVA — Repeated measures ANOVA evaluated change in outcome variables across the study time points

4. Secondary Outcome: Measure Reproductive Concerns After Cancer (RCAC) Scale
Description: The Reproductive Concerns After Cancer (RCAC) Scale is a validated survey of cancer survivors' fertility and health concerns. The survey has 18 questions, answered on a 5-point scale ranging from "strongly disagree" (1) to "strongly agree" (5). Total scores range from 18 to 90, with higher scores indicating greater distress (worse outcome).
Time Frame: Baseline, 1 month, 3 months
Population: Participants with available data at each respective timepoint
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Online Decision Aid
Number analyzed (Participants) | 98
score on a scale
  Baseline | 64.14 (11.03)
  1 month: number analyzed (Participants) | 78
  1 month | 61.55 (12.30)
  3 months: number analyzed (Participants) | 55
  3 months | 60.94 (11.19)
Statistical Analysis 1: Comparison: Online Decision Aid; Test type: Other; p = 0.10, ANOVA — Repeated measures ANOVA evaluated change in outcome variables across the study time points

5. Secondary Outcome: Measure Impact of Events Scale-Revised (IES-R)
Description: Impact of Events Scale-Revised (IES-R) is a validated measure of distress in reaction to negative life events that has been adapted to measure current subjective distress related to infertility risk. The survey has 15 questions, intended to collect the participant's assessment of intrusive thoughts (7 questions) and effortful avoidance of reminders about a distressing event (8 questions). The questions are answered on a 5-point scale ranging from "not at all" (1) to "extremely" (5). Mean scores range from 15 to 75, with higher scores indicating greater distress (worse outcome).
Time Frame: Baseline, 1 month, 3 month
Population: Participants with available data at each respective timepoint
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Online Decision Aid
Number analyzed (Participants) | 98
score on a scale
  Baseline | 1.34 (1.04)
  1 month: number analyzed (Participants) | 78
  1 month | 1.10 (.91)
  3 months: number analyzed (Participants) | 55
  3 months | 1.03 (.92)
Statistical Analysis 1: Comparison: Online Decision Aid; Test type: Other; p = .01, ANOVA — Repeated measures ANOVA evaluated change in outcome variables across the study time points

6. Secondary Outcome: Measure PROMIS Self-Efficacy (PROMIS-SE) - General Self-Efficacy Subscale
Description: The PROMIS Self-Efficacy - General Self Efficacy subscale measures the degree to which people feel confident in managing various situations, problems, and events. The survey has 4 questions intended to collect the participant's assessment of general self-efficacy The questions are answered on a 5 point scale ranging from "I am not at all confident" (1) to "I am very confident" (5).
Time Frame: Baseline, 1 month, 3 months
Population: Participants with available data at each respective timepoint
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Online Decision Aid
Number analyzed (Participants) | 98
score on a scale
  Baseline | 3.83 (0.87)
  1 month: number analyzed (Participants) | 78
  1 month | 3.91 (0.88)
  3 months: number analyzed (Participants) | 55
  3 months | 3.89 (0.75)
Statistical Analysis 1: Comparison: Online Decision Aid; Test type: Other; p = 0.59, ANOVA — Repeated measures ANOVA evaluated change in outcome variables across the study time points

7. Secondary Outcome: Measure PROMIS Self-Efficacy (PROMIS-SE) - Managing Fertility/Family-Building Issues Subscale
Description: The PROMIS Self-Efficacy - General Self-Efficacy subscale measures the degree to which people feel confident in managing various situations, problems, and events and confidence in managing difficult emotions. Questions were adapted to assess self-efficacy in managing fertility and family-building issues. The survey has 4 questions, intended to collect the participant's assessment of self-efficacy for managing fertility/family-building issues. The questions are answered on a 5 point scale ranging from "I am not at all confident" (1) to "I am very confident" (5).
Time Frame: Baseline, 1 month, 3 months
Population: Participants with available data at each respective timepoint
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Online Decision Aid
Number analyzed (Participants) | 98
score on a scale
  Baseline | 2.95 (1.07)
  1 month: number analyzed (Participants) | 78
  1 month | 3.31 (0.94)
  3 months: number analyzed (Participants) | 55
  3 months | 3.26 (0.10)
Statistical Analysis 1: Comparison: Online Decision Aid; Test type: Other; p = 0.02, ANOVA — Repeated measures ANOVA evaluated change in outcome variables across the study time points

8. Secondary Outcome: Measure PROMIS Self-Efficacy (PROMIS-SE) - Managing Difficult Emotions Subscale
Description: The PROMIS Self-Efficacy - Managing Difficult Emotions subscale measures the degree to which people feel confident in managing difficult emotions. The survey has 4 questions, intended to collect the participant's assessment of self-efficacy for managing difficult emotions. The questions are answered on a 5 point scale ranging from "I am not at all confident" (1) to "I am very confident" (5).
Time Frame: Baseline, 1 month, 3 months
Population: Participants with available data at each respective timepoint
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Online Decision Aid
Number analyzed (Participants) | 98
score on a scale
  Baseline | 3.23 (0.95)
  1 month: number analyzed (Participants) | 78
  1 month | 3.32 (0.90)
  3 months: number analyzed (Participants) | 55
  3 months | 3.27 (0.94)
Statistical Analysis 1: Comparison: Online Decision Aid; Test type: Other; p = 0.52, ANOVA — Repeated measures ANOVA evaluated change in outcome variables across the study time points

9. Secondary Outcome: Measure PROMIS Self-Efficacy (PROMIS-SE) - Managing Difficult Emotions Related to Fertility/Family-Building Subscale
Description: The PROMIS Self-Efficacy - Managing Difficult Emotions subscale measures the degree to which people feel confident in managing difficult emotions. Questions were adapted to assess self-efficacy in managing emotions related to fertility and family-building. The survey has 4 questions, intended to collect the participant's assessment of self-efficacy for managing difficult emotions related to fertility/family-building. The questions are answered on a 5 point scale ranging from "I am not at all confident" (1) to "I am very confident" (5).
Time Frame: Baseline, 1 month, 3 months
Population: Participants with available data at each respective timepoint
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Online Decision Aid
Number analyzed (Participants) | 98
score on a scale
  Baseline | 2.70 (0.93)
  1 month: number analyzed (Participants) | 78
  1 month | 2.92 (1.05)
  3 months: number analyzed (Participants) | 55
  3 months | 2.92 (1.05)
Statistical Analysis 1: Comparison: Online Decision Aid; Test type: Other; p = 0.08, ANOVA — Repeated measures ANOVA evaluated change in outcome variables across the study time points

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Online Decision Aid
All-Cause Mortality (participants affected / at risk) | 0/98
Serious Adverse Events (participants affected / at risk) | 0/98
Other Adverse Events (participants affected / at risk) | 0/98

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-10-06): https://cdn.clinicaltrials.gov/large-docs/37/NCT04059237/Prot_SAP_001.pdf
  • Informed Consent Form (2021-02-08): https://cdn.clinicaltrials.gov/large-docs/37/NCT04059237/ICF_000.pdf